CLINICAL TRIAL: NCT05654701
Title: Expanded Access Program of Palopegteriparatide in Patients With Hypoparathyroidism
Status: Approved for marketing | Type: Expanded Access
Sponsor: Ascendis Pharma Bone Diseases A/S (Industry)
Responsible Party: Sponsor
Organization: Ascendis Pharma A/S (Industry)
Other Study IDs: ASNDMAP001
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Hypoparathyroidism
Keywords: Hypoparathyroidism; Parathyroid Hormone; TransCon PTH; PTH(1-34); Expanded Access
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Palopegteriparatide (TransCon PTH) — The investigational drug Palopegteriparatide (TransCon PTH) is supplied as a solution with a concentration of 0.3 mg PTH(1-34)/mL in a single-patient-use prefilled pen intended for subcutaneous injection.

SUMMARY:
To provide palopegteriparatide (TransCon PTH), an investigational parathyroid hormone (PTH) replacement therapy in an expanded access setting for adult patients with hypoparathyroidism who have previously received PTH-treatment, who meet the eligibility criteria for this protocol as described below and have a clear unmet medical need that cannot be adequately treated by a commercial product or a clinical trial.

DETAILED DESCRIPTION:
This is an expanded access program for eligible participants who previously received PTH treatment and who are ineligible for an ongoing TransCon PTH clinical trial. The treating physician/investigator contacts Ascendis Pharma when, based on their medical opinion, a patient meets the criteria for inclusion in the expanded access program.

Participants will start with a fixed dose of study drug and will be individually and progressively titrated to an optimal dose based on serum calcium levels, followed by an individualized dosing period until palopegteriparatide is commercially available to the participant. For patients taking conventional therapy with calcium and or active forms of vitamin D, these therapies will be reduced in dose and/or discontinued during titration of palopegteriparatide.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypoparathyroidism.
* Patients with previous PTH-treatment experience.
* Serum albumin-adjusted calcium level ≥7.8 mg/dL and 25(OH) vitamin D in the normal range within 2 weeks before first dose.
* Body mass index (BMI) 17 - 40 kg/m2.
* Be willing and able to give written informed consent by signing an Institutional Review Board (IRB)-approved Informed Consent Form (ICF).

Exclusion Criteria:

* Diagnosis of pseudohypoparathyroidism.
* Currently enrolled in an investigational drug or device study or has used an investigational drug or device within 30 days or 5 half-lives (whichever is longer) of Day 1.
* Severe renal impairment (estimated glomerular filtration rate <30 mL/min/1.73m2).
* Increased risk for osteosarcoma, such as those with Paget's disease of bone or unexplained elevations of alkaline phosphatase, hereditary disorders predisposing to osteosarcoma, or with a prior history of substantial external beam or implant radiation therapy involving the skeleton
* Active malignancy within past 2 years excluding successfully resected thyroid carcinoma and non-melanoma skin cancer.
* Severe or decompensated cardiac disease within 26 weeks, including but not limited to class IV or Stage D heart failure, unstable angina, myocardial infarction or uncontrolled arrhythmias.
* Pregnant or lactating females, or females intending to become pregnant.
* Known allergy and/or sensitivity to palopegteriparatide or its excipients or prior PTH therapy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult